CLINICAL TRIAL: NCT07303374
Title: Supra-Implant Complex Stability Following Flapless Immediate Implant Placement With Socket Shield Technique Versus Connective Tissue Graft in Anterior Maxilla 1-Year Randomized Clinical Trial
Brief Title: Flapless Immediate Implant Placement With Socket Shield Technique Versus Connective Tissue Graft in Anterior Maxilla
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Dental Contiuing Education (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDCE-38122025
Record Dates: First submitted 2025-12-08; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Immediate Dental Implant Placement; Connective Tissue Graft; Socket Shield Technique
Keywords: Socket Shield; Connective tissue graft

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated into two equal groups. The test group will undergo immediate implant placement combined with the socket shield technique and a customized healing abutment, whereas the control group will receive immediate implant placement with connective tissue grafting and a customized healing abutment. A pilot surgical guide will be used for both groups. The primary outcome measure will be labio-palatal ridge dimension changes changes. Secondary outcome measures included labial soft-tissue volumetric changes, bone formation labial to the implant, vertical bone level changes and pink esthetic score. All outcomes will be evaluated after a 12-month follow-up period.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IIP+ Socket sheild (Experimental): The socket shield technique, which preserves a labial root fragment to maintain periodontal ligament support
  Interventions: Procedure: IIP+Socket Shield
- IIP+CTG (Active Comparator): connective tissue grafting which increases soft-tissue volume
  Interventions: Procedure: IIP+CTG

INTERVENTIONS:
Procedure: IIP+Socket Shield — The socket shield technique, which preserves a labial root fragment to maintain periodontal ligament support.
  Arms: IIP+ Socket sheild
Procedure: IIP+CTG — connective tissue grafting which increases soft-tissue volume
  Arms: IIP+CTG

SUMMARY:
The present study aims to compare the dimensional stability of the supra-implant complex following flapless immediate implant placement using two socket management approaches: the connective tissue graft and the socket shield technique. Three-dimensional volumetric analysis and cone-beam computed tomography (CBCT) will be employed to assess and quantify changes in soft and hard tissue thickness and height surrounding the implant site.

DETAILED DESCRIPTION:
The current study will include 28 non-restorable single maxillary anterior teeth indicated for extraction. Patients will be randomly allocated into two equal groups. The test group will undergo immediate implant placement combined with the socket shield technique and a customized healing abutment, whereas the control group will receive immediate implant placement with connective tissue grafting and a customized healing abutment. A pilot surgical guide will be used for both groups. The primary outcome measure will be labio-palatal ridge dimension changes changes. Secondary outcome measures included labial soft-tissue volumetric changes, bone formation labial to the implant, vertical bone level changes and pink esthetic score. All outcomes will be evaluated after a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Initial intact thick gingival biotype
* 2 mm band of keratinized tissue,
* Thin intact labial bone plate (< 1mm)
* Good apical bone for primary stability
* Patients who had provided an informed consent.

Exclusion Criteria:

* Immediate implants with bone grafts or guided bone regeneration procedures
* Uncontrolled diabetes mellitus
* Patients taking IV bisphosphonates for treatment of osteoporosis
* Patients with active infection related at the site of implant
* Patients with untreated active periodontal diseases.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Soft tissue Volume gain/loss | one year
  The volumetric analysis in this clinical trial will be performed to obtain profilometric measurements. intraoral scans will be taken at baseline, 6- and 12-month post-operative for each patient. The best-fit algorithm will be used to superimpose digital surface models, when comparing each area of interest (AOI) throughout out the follow up period. Unchanged neighboring teeth surfaces will be used as a reference for proper superimposition. In each patient, the AOI will be kept constant for all pairwise comparisons. The volumetric analysis software will calculate the overall buccal soft tissue volume loss/gain (mm3) within the AOI for each patient.

SECONDARY OUTCOMES:
Mid-facial gingival margin level | 12 months
  linear change of the Mid-facial gingival margin pre- and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Nael Adel Mina, Masters, Principal Investigator — International Dental Contiuing Education
Locations (1):
- International Dental contiuing education, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No